CLINICAL TRIAL: NCT05372042
Title: Testing the Efficacy of a CBT-enhanced Text Message Intervention to Reduce Symptom Burden in Individuals With Post-traumatic Stress Disorder Symptoms and Co-occurring Hazardous Drinking
Brief Title: CBT Texts for PTSD & Hazardous Drinking (Project Better)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kristen Lindgren, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00013533; 1R01AA028776-01A1 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Posttraumatic Stress Disorder; Alcohol Use
Keywords: hazardous drinking; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will receive text messages 3 days a week for a 4 week period. To keep text messages within the length of standard SMS limits (160 characters), each day's message will be sent in the form of two brief texts (each will be 160 characters or less). The content of the text messages will vary as a function of condition. Participants will be assigned to CBT text messages plus one of six combinations of framing (3: loss vs. gain vs. no framing) and mindsets (2: growth vs reminder) texts. The combination that consists of no framing and simple reminder is an active comparator as it is the version of CBT text messages closest to what has been tested previously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Loss Framing + Growth Mindset (Experimental): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that is framed with toward preventing future losses from trauma exposure, and day 3 will have a reminder that aims to instill a growth mindset about using the skill.
  Interventions: Behavioral: CBT Text Messages
- Loss Framing + Simple Reminder (Experimental): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that is framed with toward prevent future losses from trauma exposure, and day 3 will have a simple reminder to use the skill.
  Interventions: Behavioral: CBT Text Messages
- Gain Framing + Growth Mindset (Experimental): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that is framed with toward future benefits from doing so, and day 3 will have a reminder that aims to instill a growth mindset about using the skill.
  Interventions: Behavioral: CBT Text Messages
- Gain Framing + Simple Reminder (Experimental): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that is framed with toward future benefits from doing so, and day 3 will have a simple reminder to use the skill.
  Interventions: Behavioral: CBT Text Messages
- No Framing + Growth Mindset (Experimental): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that has no framing, and day 3 will have a reminder that aims to instill a growth mindset about using the skill.
  Interventions: Behavioral: CBT Text Messages
- No Framing + Simple Reminder (Active Comparator): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about CBT skill, day 2 will be a remainder to use the skill that has no framing, and day 3 will have a simple reminder to use the skill.
  Interventions: Behavioral: CBT Text Messages

INTERVENTIONS:
Behavioral: CBT Text Messages — CBT skills based text messages delivered 3x per week for four weeks

SUMMARY:
The research study seeks to refine and test a brief, self-directed, intervention for individuals from the general public with PTSD and co-occurring HD that can be delivered via text-messaging. This application seeks to refine the intervention further by testing whether theoretically-driven, evidence-based strategies from basic cognitive psychology (message framing) and social psychology (facilitating growth mindsets) result in better outcomes for PTSD symptoms and HD by addressing pilot participant feedback related to avoidance and motivation.

DETAILED DESCRIPTION:
This study will refine a previously piloted text message intervention by integrating and testing the efficacy of behavioral nudge and psychologically-wise intervention techniques when added to CBT text messages for reducing hazardous drinking (HD) and PTSD symptoms.The enhancements will be tested in a fully crossed 3 (message framing: avoid losses vs. maximize gains vs. no framing) x 2 (mindsets: facilitate growth mindset reminder vs. simple reminder to use skills) factorial design to identify the most effective combination of text messages. A sample of 500 participants with DSM-5 Criterion A trauma exposure, PTSD symptoms, and HD will be enrolled and randomized to condition. Baseline, immediate post-, 1-, and 3-month assessments will capture change in primary outcomes (PTSD, hazardous drinking).

Trauma exposure and PTSD symptoms will be assessed using the Posttraumatic Stress Disorder Checklist, Civilian Version DSM-5 with the Life Events Checklist (PCL-5 and LEC).

HD will be assessed via a set of measures that provide a detailed picture of drinking patterns. First, two questions will ask about heavy episodic drinking (HED: 4/5 or more drinks per single occasion for men/women) episodes, assessing both frequency over the lifetime and frequency over the last month. Typical weekly alcohol consumption will also be assessed using the Daily Drinking Questionnaire (DDQ). Negative alcohol-related consequences will be assessed via the Short Index of Problems (SIP).

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Currently resides in WA State
3. Fluent in English
4. Reports at least one DSM-5 traumatic event that occurred 1+ months ago
5. Current PTSD severity of 33+ on the PCL-5
6. Current hazardous alcohol use (2+ heavy episodic drinking occasions [4+ drinks on one occasion for women, 5+ drinks on one occasion for men] in past month, 1+ negative consequences related to alcohol use)
7. Owns a functioning cellular phone
8. Is willing to receive weekly study text messages for 4 consecutive weeks
9. Is willing to provide contact information including phone number (for text messages and reminders), email (reminders), and mailing address (payment)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Lindgren, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2,751 completed the screening survey, and 1,397 of them were not eligible. Among 1,354 participants who were eligible for the verification call, 628 were excluded prior to verification call due to suspected fraud, missing contact information, etc. and 162 did not show up/declined participation. Among 564 participants who were sent baseline survey, 45 never completed baseline and 14 were identified as fraudulent upon review. 505 completed baseline/enrolled and were randomized.
Period: Post Intervention
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Started | 84 | 83 | 86 | 85 | 85 | 82
Completed | 78 | 78 | 76 | 79 | 80 | 78
Not Completed | 6 | 5 | 10 | 6 | 5 | 4
Period: 1-Month Follow Up
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Started | 84 | 83 | 86 | 85 | 85 | 82
Completed | 77 | 78 | 74 | 82 | 80 | 79
Not Completed | 7 | 5 | 12 | 3 | 5 | 3
Period: 3-Month Follow Up
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Started | 84 | 83 | 86 | 85 | 85 | 82
Completed | 73 | 75 | 73 | 82 | 78 | 71
Not Completed | 11 | 8 | 13 | 3 | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder | Total
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.45 (10.98) | 38.06 (12.04) | 36.83 (10.7) | 35.99 (11.05) | 34.47 (10.19) | 35.82 (11.17) | 36.27 (11.03)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17 | 15 | 18 | 16 | 16 | 17 | 99
  Female | 55 | 60 | 59 | 61 | 63 | 62 | 360
  Transgender | 2 | 1 | 2 | 4 | 2 | 1 | 12
  Another identity | 10 | 7 | 7 | 4 | 4 | 2 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 7 | 12 | 9 | 12 | 56
  Not Hispanic or Latino | 70 | 71 | 75 | 72 | 76 | 69 | 433
  Unknown or Not Reported | 4 | 6 | 4 | 1 | 0 | 1 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 2 | 4 | 2 | 13
  Asian | 4 | 2 | 2 | 6 | 4 | 2 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 2 | 4 | 4 | 18
  White | 64 | 64 | 69 | 61 | 59 | 60 | 377
  More than one race | 12 | 9 | 7 | 14 | 10 | 10 | 62
  Unknown or Not Reported | 0 | 2 | 5 | 0 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Heavy Episodic Drinking
Description: Heavy Episodic Drinking (HED) assesses the quantity of heavy drinking episodes (i.e., >4/5 drinks per occasion for women/men, based on the National Institute of Alcohol Abuse and Alcoholism's definition) over the last month. It is administered at pre-intervention (baseline), post-intervention (week 4), 1 month follow up (week 8), and 3 month follow up (week 16). The range of the scale is 0-10 (count of the number of heavy drinking episodes in the last month); 10 is described as 10 or more heavy drinking episodes. Higher scores represent a greater number of heavy drinking episodes.
Time Frame: Baseline, 4 weeks, 8 weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: number of heavy drinking episodes
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
number of heavy drinking episodes
  Timepoint: Pre-intervention (Baseline) | 6.19 (3.03) | 6.00 (3.15) | 5.85 (3.20) | 6.69 (3.12) | 6.02 (3.12) | 6.33 (3.22)
  Timepoint: Post-intervention (Week 4) | 3.71 (3.40) | 4.58 (3.73) | 3.63 (3.45) | 4.52 (3.47) | 3.48 (3.43) | 4.03 (3.44)
  Timepoint: Month 1 follow-up (Week 8) | 3.27 (3.50) | 3.82 (3.71) | 3.32 (3.27) | 3.48 (3.61) | 3.01 (3.38) | 2.96 (3.31)
  Timepoint: Month 3 follow-up (Week 16) | 2.53 (2.98) | 3.61 (3.75) | 3.18 (3.40) | 3.65 (3.70) | 3.04 (3.33) | 2.33 (3.01)

2. Primary Outcome: Posttraumatic Stress Disorder (PTSD)
Description: The Posttraumatic Stress Disorder Checklist for the 5th Edition of Diagnostic and Statistical Manual of Mental Disorders (PCL-5) assesses the severity of symptoms of posttraumatic stress disorder (PTSD) as defined by the 5th Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and is administered at pre-intervention (baseline), post-intervention (week 4), 1 month follow up (week 8), and 3 month follow up (week 16) to assess change in PTSD symptoms. The range of the scale is 0-80. Higher scores represent more severe PTSD symptoms.
Time Frame: Baseline, 4 weeks, 8 weeks, and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline) | 51.83 (11.43) | 49.99 (11.97) | 50.66 (11.43) | 51.67 (11.87) | 51.66 (11.44) | 51.33 (11.95)
  Timepoint: Post-intervention (Week 4) | 39.72 (15.23) | 38.85 (15.75) | 38.78 (14.30) | 39.38 (15.91) | 39.40 (14.91) | 39.06 (15.72)
  Timepoint: Month 1 follow-up (Week 8) | 34.19 (14.87) | 37.73 (14.90) | 38.46 (14.39) | 37.18 (15.40) | 35.83 (16.27) | 35.14 (14.23)
  Timepoint: Month 3 follow-up (Week 16) | 33.72 (15.34) | 34.64 (18.60) | 36.53 (15.27) | 36.61 (15.36) | 34.23 (16.36) | 31.51 (16.79)

3. Primary Outcome: Typical Weekly Alcohol Consumption
Description: The Daily Drinking Questionnaire (DDQ) assesses the number of standard drinks consumed each day of a typical week over the last month and is administered at pre-intervention (baseline), post-intervention (week 4), 1 month follow up (week 8), and 3 month follow up (week 16). The range for the scale to report drinks consumed each day is 0-25. Each day's score for the week is summed to created a total number of drinks consumed per week; the count of drinks consumed per week ranges from 0 to 175. Higher scores representing greater number of drinks consumed during a typical week.
Time Frame: Baseline, 4 weeks, 8 weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: number of standard drinks per week
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
number of standard drinks per week
  Timepoint: Pre-intervention (Baseline) | 23.96 (22.19) | 26.00 (18.50) | 26.00 (26.01) | 26.15 (22.98) | 23.68 (20.97) | 25.63 (20.80)
  Timepoint: Post-intervention (Week 4) | 16.65 (19.06) | 21.49 (19.47) | 19.72 (18.91) | 18.67 (13.90) | 18.20 (19.71) | 17.96 (16.46)
  Timepoint: Month 1 follow-up (Week 8) | 14.85 (18.24) | 17.24 (16.85) | 16.46 (20.16) | 16.48 (15.21) | 15.89 (23.41) | 14.79 (16.57)
  Timepoint: Month 3 follow-up (Week 16) | 11.80 (12.86) | 17.88 (22.83) | 17.05 (23.15) | 16.24 (17.60) | 14.46 (23.58) | 11.47 (13.78)

4. Primary Outcome: Alcohol Use Consequences
Description: The Short Index of Problems (SIP) assesses the negative consequences from alcohol consumption over the last month and is administered at pre-intervention (baseline), post-intervention (week 4), 1 month follow up (week 8), and 3 month follow up (week 16). The range for the scale is 0-15 and higher scores represent a greater number of alcohol-related consequences.
Time Frame: Baseline, 4 weeks, 8 weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline) | 8.99 (3.65) | 9.00 (3.65) | 8.22 (4.07) | 9.02 (3.87) | 8.33 (4.06) | 9.28 (3.74)
  Timepoint: Post-intervention (Week 4) | 5.87 (3.90) | 6.54 (4.15) | 5.54 (4.33) | 6.14 (4.44) | 5.16 (4.31) | 5.83 (4.34)
  Timepoint: Month 1 follow-up (Week 8) | 4.68 (3.92) | 5.99 (5.10) | 4.84 (4.59) | 4.95 (4.55) | 4.76 (4.82) | 5.09 (4.72)
  Timepoint: Month 3 follow-up (Week 16) | 4.65 (4.41) | 5.06 (5.07) | 4.55 (4.76) | 4.83 (4.73) | 4.55 (5.05) | 3.49 (4.24)

5. Secondary Outcome: Risk of Alcohol Use Disorder (AUD)
Description: The Alcohol Use Disorders Identification Test (AUDIT) assesses problem drinking and likely diagnosis of an alcohol use disorder over the last 12 months and is administered at pre-intervention (baseline) and 3 month follow up (week 16). The total range of scores is 0-40 and higher scores represent greater risks of having an alcohol use disorder.
Time Frame: Baseline,16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline) | 18.29 (7.35) | 18.49 (7.02) | 18.17 (8.35) | 18.89 (8.38) | 17.72 (9.01) | 18.54 (7.18)
  Timepoint: Month 3 follow-up (Week 16) | 12.93 (7.26) | 15.63 (8.06) | 14.12 (8.06) | 15.21 (8.78) | 14.19 (9.43) | 13.23 (7.82)

6. Secondary Outcome: Depression, Anxiety, and Stress Scale
Description: The Depression Anxiety Stress Scale (DASS-21) assesses the general psychopathology symptoms over the last month and is administered at pre-intervention (baseline), 1 month follow up (week 8), and 3 month follow up (week 16). It has 3 subscales; two of which (anxiety and depression subscales) are outcomes for this study. The total range of scores of the anxiety subscale of the DASS-21 is 0-21 and higher scores indicate more severe symptoms. The total range of scores of the depression subscale of the DASS-21 is 0-21 and higher scores indicate more severe symptoms.
Time Frame: Baseline, 8 weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline), Depression | 11.15 (4.67) | 12.12 (4.89) | 12.13 (4.87) | 12.44 (4.97) | 11.79 (4.95) | 11.59 (4.69)
  Timepoint: Month 1 follow-up (Week 8), Depression | 9.40 (5.15) | 9.69 (5.46) | 10.73 (5.42) | 9.40 (5.53) | 9.61 (6.03) | 8.98 (5.55)
  Timepoint: Month 3 follow-up (Week 16), Depression | 8.93 (5.34) | 9.16 (6.25) | 10.22 (5.70) | 8.95 (5.65) | 8.96 (5.61) | 8.55 (5.12)
  Timepoint: Pre-intervention (Baseline), Anxiety | 7.92 (3.89) | 8.37 (4.74) | 8.70 (4.04) | 9.33 (3.96) | 9.05 (4.29) | 8.45 (4.27)
  Timepoint: Month 1 follow-up (Week 8), Anxiety | 6.88 (3.86) | 6.83 (4.01) | 7.14 (4.49) | 7.15 (4.25) | 6.85 (4.47) | 5.90 (4.20)
  Timepoint: Month 3 follow-up (Week 16), Anxiety | 7.00 (4.64) | 6.26 (4.76) | 6.64 (4.74) | 7.24 (4.82) | 6.27 (4.02) | 6.00 (4.08)

7. Secondary Outcome: Treatment Seeking
Description: The Treatment Services Received (TSR) assesses the types of mental health and addictions treatments that individuals (e.g., inpatient, outpatient, 12-step, etc) received since enrolling in the study and is administered at 3 month follow up (week 16). Twelve types of treatment are listed and counted to calculate the number of types of treatment that individuals received over the 16-week study period. The minimum possible score is 0 (no services received) and the maximum is 12 types of treatment. Higher numbers indicate receiving more types of treatment.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: unique mental health treatments
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
unique mental health treatments | 0.61 (1.03) | 0.49 (0.80) | 0.43 (0.73) | 0.82 (1.19) | 0.47 (0.92) | 0.42 (0.88)

8. Secondary Outcome: Drug Use
Description: The Customary Drinking and Drug Use Record (CDDR) assesses comprehensive substance use, other than alcohol, over the last 3 months and is administered at pre-intervention (baseline) and 3 month follow up (week 16). The total range of scores is 0-12 and higher scores indicate more drug use.
Time Frame: Baseline,16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline) | 3.82 (2.60) | 4.24 (3.12) | 3.51 (2.50) | 3.61 (2.74) | 3.79 (3.17) | 4.05 (3.11)
  Timepoint: Month 3 follow-up (Week 16) | 2.18 (2.04) | 2.00 (1.67) | 2.00 (2.25) | 1.87 (1.94) | 1.86 (2.12) | 1.81 (2.03)

9. Secondary Outcome: Drug Use Problems
Description: The Drug Abuse Screening Test (DAST-10) assesses the problems related to other substance use and likely drug use disorder diagnosis over the last 12 months and is administered at pre-intervention (baseline) and 3 month follow up (week 16). The total range of scores is 0-10 and higher scores indicate more substance use-related problems and likely drug use disorder diagnosis.
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
Number analyzed (Participants) | 84 | 83 | 86 | 85 | 85 | 82
score on a scale
  Timepoint: Pre-intervention (Baseline) | 3.24 (2.66) | 3.60 (3.23) | 2.86 (2.64) | 3.06 (3.08) | 2.87 (3.01) | 3.48 (2.95)
  Timepoint: Month 3 follow-up (Week 16) | 2.32 (2.48) | 2.38 (2.68) | 1.67 (2.35) | 2.36 (3.04) | 1.79 (2.44) | 1.81 (2.57)

ADVERSE EVENTS:
Time Frame: The study collected adverse event data for participants for 4 month (16 weeks) following baseline. Adverse event event information was collected through study completion.
Description: This is study is a brief text message psychosocial intervention for individuals with PTSD symptoms and co-occurring hazardous drinking. Risks for participation were expected to be potential discomfort with answering questions about mental health and substance use. No serious adverse events were anticipated, and the study was judged to be minimal risk by the IRB.
Arm/Group | Loss Framing + Growth Mindset | Loss Framing + Simple Reminder | Gain Framing + Growth Mindset | Gain Framing + Simple Reminder | No Framing + Growth Mindset | No Framing + Simple Reminder
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83 | 0/86 | 0/85 | 0/85 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83 | 0/86 | 0/85 | 0/85 | 0/82
Other Adverse Events (participants affected / at risk) | 0/84 | 0/83 | 0/86 | 0/85 | 0/85 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT05372042/Prot_SAP_000.pdf